CLINICAL TRIAL: NCT03742635
Title: Feasibility and Reliability of Applying Prechtl's Assessment of General Movements for Preterm Infants Through Telemedicine
Brief Title: Applying Prechtl's Assessment of General Movements for Preterm Infants Through Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1288981
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Infant, Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Conduct General Movements Assessments (GMA) both in-person/via telemedicine ("real-time") and through recordings (standard of care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GMA Assessment (Experimental): Conduct General Movements Assessment (GMA) in-person/via-telemedicne ("real-time") and recorded (standard of care)
  Interventions: Other: General Movements Assessment

INTERVENTIONS:
Other: General Movements Assessment — Prechtl's Assessment of General Movements (GMA) is a tool used in early infancy to identify infants at high risk of cerebral palsy and neurodevelopmental impairment. General movements are complex motor patterns that involve the entire body, moving fluidly in different directions through the arms, legs, and trunk with variable speed, amplitude, force and intensity. During fetal development, spontaneously generated motor patterns, including general movements, can already be observed. The GMA is a functional assessment of the maturing nervous system that takes advantage of the fact that typically developing infants will have a progression in their general movements. This pattern is characterized by a writhing pattern in the early weeks post-term, followed by the emergence of fidgety movements at 3-5 months of age.

SUMMARY:
The investigators will implement a study to evaluate the hypothesis that applying General Movements Assessments (GMA) in a telemedicine setting with real-time scoring is feasible and comparable to scoring video recordings.

DETAILED DESCRIPTION:
The investigators hypothesize that using telemedicine to conduct the GMA will improve early identification of risk for cerebral palsy and facilitate earlier referral and access to neurodevelopmental intervention. Preterm birth results from complex interactions of biological and socioeconomic risk factors, all of which continue to influence neurodevelopmental trajectories beyond the prenatal and neonatal period. Unfortunately many of the socioeconomic factors that contribute to increased risk of prematurity are also associated with decreased likelihood to attend appointments at high risk infant follow-up (HRIF) clinics. Early intervention has been shown to be most beneficial to infants with highest social risk. Additionally, mothers living in more rural communities tend to have higher social risk. They are often younger, more likely to be a single parent, and have lower income. Helping make follow-up more accessible and convenient for families through telemedicine and at an earlier age using the GMA has the potential to improve early identification, minimize loss to follow-up and ensure prompt referral to optimize outcomes for the most vulnerable babies in this already high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants who meet the High-Risk Infant Follow Up (HRIF) Criteria (less than 32 weeks gestational age or birth weight less than 1500 grams) who are cared for at UC Davis Medical Center

Exclusion Criteria:

* Families who are non-English speakers requiring a translator
* Families who are unable to access data-capable wireless service to participate in telemedicine visits through Zoom.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Real-time versus video recording reliability | 9 months gestational age
  Intra-rater reliability of GMA (real-time versus video recording) will be assessed using the Kappa statistic.

SECONDARY OUTCOMES:
Video recording reliability | 9 months gestational age
  Inter-rater reliability of the video recording will be assessed using the Kappa statistic.
Early referral | 9 months gestational age
  Number of participants referred to targeted early intervention services, indicating early recognition of neurodevelopmental disability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No